CLINICAL TRIAL: NCT00880607
Title: The Use of Intraoperative Intrathecal Morphine Versus Epidural Extended Release Morphine for Postoperative Pain Control in Pediatric Patients Undergoing Posterior Spinal Fusion
Brief Title: Intrathecal Morphine Versus Epidural Extended Release Morphine for Pediatric Patients Undergoing Spinal Fusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-0721; Seed grant UCHSC (Other: University of Colorado Department of Anesthesiology)
Record Dates: First submitted 2009-04-10; First posted 2009-04-14 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Pain Management; Spinal Fusion; Scoliosis
Keywords: Pain; Pediatric; Spinal Fusion; pain management
MeSH Terms: conditions — Agnosia; Scoliosis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intrathecal morphine (Active Comparator): Receives a single dose of intrathecal morphine
  Interventions: Drug: Intrathecal morphine
- Extended Release Epidural Morphine (Experimental): Receives DepoDur extended release epidural morphine for pain management
  Interventions: Drug: Extended Release Epidural Morphine

INTERVENTIONS:
Drug: Intrathecal morphine — Morphine injection is a systemic narcotic analgesic for administration by the intravenous, epidural or intrathecal routes. It is used for the management of pain.
  Other Names: IT Morphine
  Arms: Intrathecal morphine
Drug: Extended Release Epidural Morphine — DepoDur™ is a preparation of extended release lipid encapsulated morphine and is used specifically for epidural injection, outside the spinal fluid, for postoperative pain. This study is a prospective randomized double-blinded trial examining the effectiveness of single dose intrathecal morphine versus single dose extended release epidural morphine for postoperative pain control in pediatric posterior spinal fusion patients.
  Other Names: EREM; DepoDur
  Arms: Extended Release Epidural Morphine

SUMMARY:
This study plans to learn more about preventing pain in children who are having posterior spinal fusion surgery using two different kinds of morphine (a pain medicine). Also, this study plans to learn about individual differences in the how the different kinds of morphine work in children.

Subjects are being asked to be in this research study because they are having spinal fusion surgery, will have pain some of the time and will be getting morphine during and after surgery to help control their pain.

DETAILED DESCRIPTION:
Up to 80 people from Denver will participate in the study. Subjects will be randomized to receive one of two possible medications during surgery to help with pain after surgery. After they go to sleep for surgery the anesthesiologist will give them either (1) a single injection of morphine into the spinal fluid in the lower back, or (2) a single injection of extended-release morphine into the epidural space (just outside the spinal fluid) in the lower back.

The usual care for patients having this surgery is a single injection of morphine into the spinal fluid in the lower back. If randomized to group (1), subjects will receive the usual care for pain control. If subjects are randomized to group (2), they will receive a single injection of extended-release morphine into the epidural space.

During surgery, a small blood sample (1 teaspoon or less) will be collected to analyze specific DNA sequences that are involved in individual responses to morphine for pain control. The blood sample will be destroyed after 24 months.

After surgery, subjects will have IV pain medication through a patient-controlled analgesia (PCA) machine. Subjects will be shown how to work the PCA so they can get the pain medicine when they need it. A research nurse will check in frequently to ask how much pain is occurring following the surgery and any side effects that may arise from the study medicine.

Subjects will be in this study up to 60 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females, 8 to17 years old undergoing posterior spinal fusion for idiopathic scoliosis.
2. Fusion of a minimum of 5, and a maximum of 13 levels, including at least L1 or lower.

Exclusion Criteria:

1. Neuromuscular scoliosis.
2. A history of documented coagulopathy or platelet count of less than 100,000 mm3.
3. A known allergy or adverse sensitivity to morphine.
4. Pulmonary hypertension or other significant respiratory problem.
5. Cognitive deficits that would impair use of PCA and/or filling out questionnaire.
6. History of sleep apnea defined by sleep study and/or need for nighttime CPAP.
7. Abnormal pain thresholds (i.e., subjects who are on significant opioids preoperatively).
8. Baseline neurologic deficits (numbness, motor deficits, or any focal neurological sign).
9. Subjects who are anticipated to remain intubated postoperatively for longer than 2 hours.
10. Need for preoperative intravenous inotropic drugs.
11. Significant metabolic, endocrine or neuropathology, cyanosis, or renal insufficiency.
12. A contraindication to dural puncture, such as raised intracranial pressure.
13. Pre-operative heparin, oral aspirin or anticoagulants.
14. Weight less than 20kg or greater than 100kg.
15. Need for Intraoperative ketamine administration.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mindy Cohen, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- The Children's Hospital- Denver, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 84 patients consented to participate. 3 patients did not start the study due to physician discretion.
Groups:
- DepoDur: Receives DepoDur extended release morphine for pain management
  DepoDur: DepoDur™ is a preparation of extended release lipid encapsulated morphine and is used specifically for epidural injection, outside the spinal fluid, for postoperative pain. This study is a prospective randomized double-blinded trial examining the effectiveness of single dose intrathecal morphine versus single dose extended release epidural morphine for postoperative pain control in pediatric posterior spinal fusion patients.
Period: Overall Study
Arm/Group | Intrathecal Morphine | DepoDur
Started | 44 | 37
Observation After Receiving Medication | 42 | 35
Completed | 37 | 34
Not Completed | 7 | 3
Not completed — Physician Decision | 2 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — surgery did not extend past L1 level | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intrathecal Morphine | DepoDur | Total
Number analyzed (Participants) | 37 | 34 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (1.9) | 14.2 (1.9) | 14.0 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 29 | 29 | 58
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 34 | 71
Weight [Mean (Standard Deviation); unit: kg] | 53.6 (12.0) | 55.2 (10.44) | 54.4 (11.20)

OUTCOME MEASURES:

1. Primary Outcome: Total IV Morphine Consumption up to 48 Hours Post Surgery
Description: Total IV morphine consumption during the first 0- 48 hours after surgery.Postoperative pain was treated with morphine PCA, ketorolac, oral oxycodone, and acetaminophen.
Time Frame: Four hour intervals for up to 48 hours
Population: Intent to treat pediatric patients between 8-17 years of age undergoing thoracolumbar posterior spinal fusion with either Intrathecal morphine versus extended-release epidural morphine for post operative pain control.
Measure: Median (95% Confidence Interval); unit: mg
Groups:
- Intrathecal Morphine: single dose of intrathecal morphine
  Intrathecal morphine: Morphine injection is a systemic narcotic analgesic for administration by the intravenous, epidural or intrathecal routes. It is used for the management of pain.
- EREM: Receives extended release epidural morphine for pain management
  DepoDur: DepoDur™ is a preparation of extended release lipid encapsulated morphine and is used specifically for epidural injection, outside the spinal fluid, for postoperative pain. This study is a prospective randomized double-blinded trial examining the effectiveness of single dose intrathecal morphine versus single dose extended release epidural morphine for postoperative pain control in pediatric posterior spinal fusion patients.
Arm/Group | Intrathecal Morphine | EREM
Number analyzed (Participants) | 37 | 34
mg | 34.0 [4.5 to 128.8] | 42.2 [5.5 to 123.0]
Statistical Analysis 1: Comparison: Intrathecal Morphine vs EREM; Test type: Other — Wilcoxon rank-sum test because the outcome variable was found to have a skewed distribution; p = .27, Wilcoxon (Mann-Whitney) — Hodges-Lehmanne estimation method; Median Difference (Final Values) = 7.7, 95% CI 2-sided [-5.8 to 21.2] — Hodges-Lehmanne estimation method

2. Secondary Outcome: Time Until First PCA Demand Request
Description: At 4-hour intervals for up to 48 hours IV PCA demands.
Time Frame: every 4 hours up to 48 hours
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Groups:
- Intrathecal Morphine: Intrathecal morphine
  Receives a single dose of intrathecal morphine
- EREM: extended-release epidural morphine is marketed as DepoDurTM which is a preservative-free sterile suspension of multivesicular liposomes (DepoFoam®) containing morphine, intended for epidural administration. DepoFoam consists of lipid-based particles containing discrete water-filled chambers dispersed through the lipid matrix. The lipids are naturally occurring substances such as phospholipids and triglycerides. The small amount of lipid is cleared rapidly in the body as the particles deliver their drug payload
Arm/Group | Intrathecal Morphine | EREM
Number analyzed (Participants) | 34 | 30
hours | 0.99 [0.7500 to 1.1500] | 0.92 [0.5833 to 1.4333]
Statistical Analysis 1: Comparison: Intrathecal Morphine vs EREM; Test type: Other — Log-rank test in Kaplan-Meier used; p = .42, Log Rank

3. Secondary Outcome: Post-operative Pain Scores
Description: Post-operative pain scores using Bieri faces scale every 4 hours up to 48 hours. Using Bieri faces pain scale. The faces show how much something can hurt. The "happy face" with a smile is no pain = 0 to faces showing more and more pain up 10. The space between two faces is scored 1, 3,5,7, or 9. to 10 (worst pain) will be used every 4 hours post-op for up to 48 hours.
  *Scores were not collected and/or included for all participants at all time points. If a patient was sleeping, there score was not recorded. If a patient completed the pain scale incorrectly (used an even number or included a range), then the data point was not included.
Time Frame: every 4 hours up to 48 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intrathecal Morphine | EREM
Number analyzed (Participants) | 37 | 34
units on a scale
  0 hours: number analyzed (Participants) | 35 | 24
  0 hours | 3.26 (0.53) | 6.69 (0.60)
  4 hours: number analyzed (Participants) | 33 | 31
  4 hours | 2.70 (0.38) | 4.03 (0.46)
  8 hours: number analyzed (Participants) | 36 | 26
  8 hours | 2.25 (0.36) | 2.88 (0.43)
  12 hours: number analyzed (Participants) | 27 | 26
  12 hours | 2.96 (0.37) | 2.19 (0.44)
  16 hours: number analyzed (Participants) | 31 | 29
  16 hours | 4.13 (0.45) | 3.03 (0.38)
  20 hours: number analyzed (Participants) | 31 | 31
  20 hours | 3.61 (0.35) | 2.80 (0.34)
  24 hours: number analyzed (Participants) | 30 | 29
  24 hours | 3.10 (0.40) | 3.17 (0.36)
  32 hours: number analyzed (Participants) | 30 | 21
  32 hours | 3.83 (0.45) | 2.81 (0.34)
  36 hours: number analyzed (Participants) | 27 | 21
  36 hours | 3.85 (0.57) | 2.86 (0.35)
  40 hours: number analyzed (Participants) | 26 | 23
  40 hours | 3.92 (0.48) | 3.09 (0.43)
  44 hours: number analyzed (Participants) | 30 | 28
  44 hours | 3.63 (0.42) | 3.10 (0.36)
  48 hours: number analyzed (Participants) | 29 | 25
  48 hours | 3.41 (0.37) | 3.77 (0.35)

4. Secondary Outcome: Adverse Opioid Effect: Nausea
Description: presence of nausea- dichotomous variable
Time Frame: every 4 hours up to 48 hours
Population: as for outcome 1
Measure: Number; unit: percentage of patients with nausea
Arm/Group | Intrathecal Morphine | EREM
Number analyzed (Participants) | 37 | 34
percentage of patients with nausea | 46 | 26
Statistical Analysis 1: Comparison: Intrathecal Morphine vs EREM; Test type: Other; p = 0.08, Chi-squared

5. Secondary Outcome: Adverse Opioid Effect: Emesis
Description: presence of emesis- dichotomous variable
Time Frame: every 4 hours up to 48 hours
Population: as for outcome 1
Measure: Number; unit: percentage of patients with emesis
Arm/Group | Intrathecal Morphine | EREM
Number analyzed (Participants) | 37 | 34
percentage of patients with emesis | 24 | 15
Statistical Analysis 1: Comparison: Intrathecal Morphine vs EREM; Test type: Other; p = 0.30, Chi-squared

6. Secondary Outcome: Adverse Opioid Effect: Pruritus
Description: presence of pruritus- dichotomous variable
Time Frame: every 4 hours up to 48 hours
Population: as for outcome 1
Measure: Number; unit: percentage of patients with pruritus
Arm/Group | Intrathecal Morphine | EREM
Number analyzed (Participants) | 37 | 34
percentage of patients with pruritus | 81 | 62
Statistical Analysis 1: Comparison: Intrathecal Morphine vs EREM; Test type: Other; p = 0.07, Chi-squared

7. Secondary Outcome: Adverse Opioid Effect: Respiratory Depression
Description: presence of respiratory depression- dichotomous variable
Time Frame: every 4 hours up to 48 hours
Population: as for outcome 1
Measure: Number; unit: % patients with respiratory depression
Arm/Group | Intrathecal Morphine | EREM
Number analyzed (Participants) | 37 | 34
% patients with respiratory depression | 24 | 15
Statistical Analysis 1: Comparison: Intrathecal Morphine vs EREM; Test type: Other; p = 0.31, Chi-squared

ADVERSE EVENTS:
Time Frame: Immediately Post Op to 48 hours after surgery
Arm/Group | Intrathecal Morphine | DepoDur
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/34
Other Adverse Events (participants affected / at risk) | 0/37 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes